CLINICAL TRIAL: NCT04595331
Title: Open Label Extension for 43USSA1812 (A Randomized, Evaluator-blinded, No-treatment Controlled, Multi-center Study to Evaluate the Effectiveness and Safety of Sculptra Aesthetic for Correction of Cheek Wrinkles)
Brief Title: Open Label Extension for 43USSA1812
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 43USSA1812ext
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cheek; Wrinkle
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: Subjects originally randomized to Control Group at baseline in the pivotal 43USSA1812 study will be offered treatment with Sculptra Aesthetic in the extension study. Subjects originally randomized to Treatment Group at baseline in the pivotal 43USSA1812 study will be continued to be followed up during the extension study without further treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group A: Sculptra Aesthetic (Experimental): Subjects in this group will be treated with Sculptra aesthetic. Subjects will be followed for up to 12 months for safety and effectiveness data collection
  Interventions: Device: Sculptra Aethestic reconsituted with 8ml Sterile Water for Injection
- Group B: No Treatment (Experimental): Subjects in this group will be followed for up to 12 months with no additional treatment for long-term safety and effectiveness data collection.
  Interventions: Device: Sculptra Aethestic reconsituted with 8ml Sterile Water for Injection

INTERVENTIONS:
Device: Sculptra Aethestic reconsituted with 8ml Sterile Water for Injection — Sculptra Aesthetic 8ml and Lidocaine treatment of cheek wrinkles

SUMMARY:
To evaluate long-term safety and effectiveness data of Sculptra Aesthetic beyond the Month 12 duration of the pivotal study 43USSA1812 (NCT04124692) to help characterize the long-term safety and effectiveness profile of the more dilute suspension.

ELIGIBILITY:
Inclusion Criteria:

1. Subject completed Month 12 of study 43USSA1812
2. Subjects willing to comply with the requirements of the extension of the study and providing a signed written informed consent.

Exclusion Criteria:

1. For subjects eligible for treatment in the extension study, the exclusion criteria for study 43USSA1812 applies.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Galderma Research Site, Scottsdale, Arizona
  - Galderma Research Site, Encino, California
  - Galderma Research Site, Redondo Beach, California
  - Galderma Research site, San Diego, California
  - Galderma Research Site, Washington D.C., District of Columbia
  - Galderma Research Site, Coral Gables, Florida
  - Galderma Research Site, Alpharetta, Georgia
  - Galderma Research Site, New Orleans, Louisiana
  - Galderma Research Site, Rockville, Maryland
  - Galderma Research Site, New York, New York
  - Galderma Research Site, Dallas, Texas
  - Galderma Research Site, Spring, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 13 sites at the United States.
Pre-assignment Details: A total of 111 participants were enrolled in this extension study upon completion of 43USSA1812 (NCT04124692) study.
Groups:
- Group A: Sculptra Aesthetic: Participants in this group were treated with Sculptra aesthetic. Participants were followed for up to 12 months for safety and effectiveness data collection in this study.
- Group B: No Treatment: Participants in this group followed for long-term safety and effectiveness with no additional treatment. Participants were followed for up to 12 months for safety and effectiveness data collection in this study.
Period: Overall Study
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Started | 39 | 72
Completed | 39 | 65
Not Completed | 0 | 7
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 5
Not completed — Medical reason | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment | Total
Number analyzed (Participants) | 39 | 72 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (7.46) | 60.8 (8.06) | 60.4 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 69 | 107
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 34 | 69 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 36 | 64 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Fitzpatrick skin type (FST) [Count of Participants; unit: Participants] — FST I: white; very fair; red or blond hair; blue eyes; freckles. always burns, never tans.
  FST II: white; fair; red or blond hair; blue, hazel or green eyes. usually burns, tans with difficulty.
  FST III: cream white; fair with any eye or hair color; very common. sometimes mild burn, gradually tans.
  FST IV: brown; typical Mediterranean Caucasian skin. rarely burns, tans with ease.
  FST V: dark brown; Middle Eastern skin types. very rarely burns, tans very easily.
  FST VI: Skin color - black. Skin Characteristics - never burns, tans very easily.
  Participants
    FST I | 1 | 3 | 4
    FST II | 14 | 18 | 32
    FST III | 16 | 36 | 52
    FST IV | 4 | 8 | 12
    FST V | 3 | 4 | 7
    FST VI | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate Based on the Blinded Evaluator's Live Assessment of the Galderma Cheek Wrinkles Scale (GCWS) at Rest
Description: Responder rate was defined as the percentage of participants with at least a 1-grade improvement from baseline on the GCWS, on both sides of the face, concurrently. GCWS is a validated 5-point scale used to assess the severity of cheek wrinkles on as scale of 0 to 4. Higher score means more severe (worse) wrinkles. The participant was to have a relaxed face during the assessment.
Time Frame: At Months 19, 21 and 24 (4 weeks is defined as one month in the study / study follow up windows for certain visits were +/- 2 weeks)
Population: The extension population included all participants entering the extension study. Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure and "number analyzed" refer to participants evaluable for this outcome at given timepoints.
  (4 weeks is defined as one month in the study / study follow up windows for certain visits were +/- 2 weeks)
Measure: Number; unit: Percentage of participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 38 | 66
Percentage of participants
  At Month 19: number analyzed (Participants) | 36 | 66
  At Month 19 | 33.3 | 84.8
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21 | 36.8 | 76.9
  At Month 24: number analyzed (Participants) | 38 | 65
  At Month 24 | 42.1 | 76.9

2. Secondary Outcome: Responder Rate Based on the Blinded Evaluator's Live Assessment of the GCWS Dynamic
Description: Responder rate was defined as the percentage of participants with at least a 1-grade improvement from baseline on the GCWS, on both sides of the face, concurrently. GCWS is a validated 5-point scale used to assess the severity of cheek wrinkles on a scale of 0 to 4. Higher score means more severe (worse) wrinkles. The participant was to have a closed maximum smile during the assessment.
Time Frame: At Months 19, 21, and 24 (4 weeks is defined as one month in the study / study follow up windows for certain visits were +/- 2 weeks)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 38 | 66
Percentage of participants
  At Month 19: number analyzed (Participants) | 36 | 66
  At Month 19 | 41.7 | 77.3
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21 | 44.7 | 75.4
  At Month 24: number analyzed (Participants) | 38 | 65
  At Month 24 | 50 | 73.8

3. Secondary Outcome: Percentage of Participants With At Least "Improved" on the Global Aesthetic Improvement Scale (GAIS) Based on the Participants Live Assessment
Description: GAIS responder rates are based on independent assessments by the participant. Responder rate was defined as the percentage of participants with at least "Improved" when compared to baseline before first treatment. The 7-graded GAIS was used by the participant to rate their aesthetic improvement of the cheek wrinkles on a scale from "Very Much Improved" to "Very Much Worse" in a live assessment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 66
Percentage of participants
  At Month 19: number analyzed (Participants) | 36 | 66
  At Month 19 | 97.2 | 97.0
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21 | 97.4 | 96.9
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24 | 92.3 | 93.8

4. Secondary Outcome: Percentage of Participants With At Least "Improved" on the GAIS Based on the Investigator Live Assessment
Description: GAIS responder rates are based on independent assessments by the investigator. Responder rate was defined as the percentage of participants with at least "Improved" when compared to baseline before first treatment. The 7-graded GAIS was used by the investigator to rate aesthetic improvement of the cheek wrinkles on a scale from "Very Much Improved" to "Very Much Worse" in a live assessment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 66
Percentage of participants
  At Month 19: number analyzed (Participants) | 36 | 66
  At Month 19 | 97.2 | 97.0
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21 | 97.4 | 96.9
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24 | 92.3 | 93.8

5. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Make You Look Younger?
Description: A 5-point subject satisfaction questionnaire with the following responses: Excellent, Very good, Good, Satisfactory, Not satisfied.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 67
Participants
  At Month 19: number analyzed (Participants) | 36 | 67
  At Month 19: Excellent | 8 | 14
  At Month 19: Very good | 8 | 14
  At Month 19: Good | 10 | 21
  At Month 19: Satisfactory | 8 | 13
  At Month 19: Not satisfied | 2 | 5
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21: Excellent | 6 | 16
  At Month 21: Very good | 12 | 13
  At Month 21: Good | 11 | 17
  At Month 21: Satisfactory | 6 | 18
  At Month 21: Not satisfied | 3 | 1
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24: Excellent | 7 | 14
  At Month 24: Very good | 14 | 12
  At Month 24: Good | 10 | 21
  At Month 24: Satisfactory | 5 | 11
  At Month 24: Not satisfied | 3 | 7

6. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Make You Feel Better About Yourself?
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 67
Participants
  At Month 19: number analyzed (Participants) | 36 | 67
  At Month 19: Excellent | 7 | 14
  At Month 19: Very Good | 9 | 18
  At Month 19: Good | 11 | 19
  At Month 19: Satisfactory | 7 | 13
  At Month 19: Not Satisfied | 2 | 3
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21: Excellent | 6 | 16
  At Month 21: Very Good | 11 | 14
  At Month 21: Good | 12 | 17
  At Month 21: Satisfactory | 7 | 15
  At Month 21: Not Satisfied | 2 | 3
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24: Excellent | 7 | 15
  At Month 24: Very Good | 17 | 13
  At Month 24: Good | 8 | 19
  At Month 24: Satisfactory | 4 | 13
  At Month 24: Not Satisfied | 3 | 5

7. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Improve Your Self-confidence?
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 67
Participants
  At Month 19: number analyzed (Participants) | 36 | 67
  At Month 19: Excellent | 5 | 14
  At Month 19: Very good | 10 | 17
  At Month 19: Good | 12 | 17
  At Month 19: Satisfactory | 7 | 16
  At Month 19: Not Satisfied | 2 | 3
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21: Excellent | 6 | 15
  At Month 21: Very good | 9 | 15
  At Month 21: Good | 12 | 16
  At Month 21: Satisfactory | 7 | 15
  At Month 21: Not Satisfied | 4 | 4
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24: Excellent | 7 | 14
  At Month 24: Very good | 14 | 12
  At Month 24: Good | 10 | 21
  At Month 24: Satisfactory | 5 | 11
  At Month 24: Not Satisfied | 3 | 7

8. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Improve Overall Satisfaction With Your Appearance?
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 67
Participants
  At Month 19: number analyzed (Participants) | 36 | 67
  At Month 19: Excellent | 4 | 16
  At Month 19: Very Good | 14 | 14
  At Month 19: Good | 9 | 20
  At Month 19: Satisfactory | 7 | 12
  At Month 19: Not Satisfied | 2 | 5
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21: Excellent | 7 | 16
  At Month 21: Very Good | 9 | 16
  At Month 21: Good | 14 | 16
  At Month 21: Satisfactory | 5 | 13
  At Month 21: Not Satisfied | 3 | 4
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24: Excellent | 7 | 15
  At Month 24: Very Good | 15 | 13
  At Month 24: Good | 10 | 20
  At Month 24: Satisfactory | 3 | 10
  At Month 24: Not Satisfied | 4 | 7

9. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Make You Look/Feel More Confident in Your Life?
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 67
Participants
  At Month 19: number analyzed (Participants) | 36 | 67
  At Month 19: Excellent | 3 | 15
  At Month 19: Very good | 12 | 14
  At Month 19: Good | 12 | 19
  At Month 19: Satisfactory | 7 | 14
  At Month 19: Not Satisfied | 2 | 5
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21: Excellent | 5 | 16
  At Month 21: Very good | 10 | 13
  At Month 21: Good | 13 | 15
  At Month 21: Satisfactory | 6 | 17
  At Month 21: Not Satisfied | 4 | 4
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24: Excellent | 7 | 13
  At Month 24: Very good | 13 | 13
  At Month 24: Good | 11 | 20
  At Month 24: Satisfactory | 5 | 15
  At Month 24: Not Satisfied | 3 | 4

10. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Make You Look the Way You Feel?
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 67
Participants
  At Month 19: number analyzed (Participants) | 36 | 67
  At Month 19: Excellent | 6 | 13
  At Month 19: Very good | 11 | 14
  At Month 19: Good | 11 | 18
  At Month 19: Satisfactory | 5 | 18
  At Month 19: Not Satisfied | 3 | 4
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21: Excellent | 4 | 16
  At Month 21: Very good | 11 | 13
  At Month 21: Good | 14 | 13
  At Month 21: Satisfactory | 5 | 18
  At Month 21: Not Satisfied | 4 | 5
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24: Excellent | 7 | 13
  At Month 24: Very good | 13 | 16
  At Month 24: Good | 11 | 16
  At Month 24: Satisfactory | 5 | 14
  At Month 24: Not Satisfied | 3 | 6

11. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Improve Your Skin Firmness?
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 67
Participants
  At Month 19: number analyzed (Participants) | 36 | 67
  At Month 19: Excellent | 9 | 14
  At Month 19: Very good | 12 | 20
  At Month 19: Good | 7 | 17
  At Month 19: Satisfactory | 5 | 12
  At Month 19: Not Satisfied | 3 | 4
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21: Excellent | 6 | 17
  At Month 21: Very good | 14 | 14
  At Month 21: Good | 10 | 17
  At Month 21: Satisfactory | 5 | 14
  At Month 21: Not Satisfied | 3 | 3
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24: Excellent | 7 | 17
  At Month 24: Very good | 14 | 10
  At Month 24: Good | 11 | 21
  At Month 24: Satisfactory | 4 | 10
  At Month 24: Not Satisfied | 3 | 7

12. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Improve Your Skin Radiance?
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 67
Participants
  At Month 19: number analyzed (Participants) | 36 | 67
  At Month 19: Excellent | 7 | 14
  At Month 19: Very good | 9 | 18
  At Month 19: Good | 11 | 19
  At Month 19: Satisfactory | 7 | 13
  At Month 19: Not Satisfied | 2 | 3
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21: Excellent | 6 | 19
  At Month 21: Very good | 12 | 12
  At Month 21: Good | 11 | 14
  At Month 21: Satisfactory | 6 | 16
  At Month 21: Not Satisfied | 3 | 4
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24: Excellent | 6 | 18
  At Month 24: Very good | 14 | 11
  At Month 24: Good | 12 | 19
  At Month 24: Satisfactory | 4 | 11
  At Month 24: Not Satisfied | 3 | 6

13. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Improve Your Skin Sagging?
Description: A 5-point subject satisfaction questionnaire with the following responses: Very Satisfied, Satisfied, Neutral, Dissatisfied, Very Dissatisfied.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 67
Participants
  At Month 19: number analyzed (Participants) | 36 | 67
  At Month 19: Excellent | 7 | 14
  At Month 19: Very good | 8 | 13
  At Month 19: Good | 13 | 17
  At Month 19: Satisfactory | 4 | 13
  At Month 19: Not Satisfied | 4 | 10
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21: Excellent | 4 | 16
  At Month 21: Very good | 13 | 16
  At Month 21: Good | 11 | 15
  At Month 21: Satisfactory | 6 | 12
  At Month 21: Not Satisfied | 4 | 6
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24: Excellent | 7 | 16
  At Month 24: Very good | 12 | 11
  At Month 24: Good | 11 | 20
  At Month 24: Satisfactory | 5 | 10
  At Month 24: Not Satisfied | 4 | 8

14. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Make Your Skin Look More Refreshed?
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 67
Participants
  At Month 19: number analyzed (Participants) | 36 | 67
  At Month 19: Excellent | 8 | 18
  At Month 19: Very good | 10 | 14
  At Month 19: Good | 10 | 13
  At Month 19: Satisfactory | 6 | 17
  At Month 19: Not satisfied | 2 | 5
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21: Excellent | 7 | 17
  At Month 21: Very good | 12 | 11
  At Month 21: Good | 10 | 19
  At Month 21: Satisfactory | 6 | 14
  At Month 21: Not satisfied | 3 | 4
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24: Excellent | 7 | 18
  At Month 24: Very good | 15 | 9
  At Month 24: Good | 9 | 20
  At Month 24: Satisfactory | 5 | 13
  At Month 24: Not satisfied | 3 | 5

15. Secondary Outcome: Subject Satisfaction: Would You Say That the Treatment Results Are Natural Looking?
Description: A 5-point subject satisfaction questionnaire with the following responses: Strongly agree, Agree, Neither agree or Disagree, Disagree, Strongly disagree.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 67
Participants
  At Month 19: number analyzed (Participants) | 36 | 67
  At Month 19: Strongly agree | 22 | 37
  At Month 19: Agree | 10 | 20
  At Month 19: Neither Agree or Disagree | 4 | 10
  At Month 19: Disagree | 0 | 0
  At Month 19: Strongly Disagree | 0 | 0
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21: Strongly agree | 21 | 35
  At Month 21: Agree | 13 | 25
  At Month 21: Neither Agree or Disagree | 4 | 5
  At Month 21: Disagree | 0 | 0
  At Month 21: Strongly Disagree | 0 | 0
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24: Strongly agree | 21 | 34
  At Month 24: Agree | 15 | 24
  At Month 24: Neither Agree or Disagree | 3 | 7
  At Month 24: Disagree | 0 | 0
  At Month 24: Strongly Disagree | 0 | 0

16. Secondary Outcome: Subject Satisfaction: Would You Say the Subtle Changes Over Time Was Worth It?
Description: as for outcome 15
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 67
Participants
  At Month 19: number analyzed (Participants) | 36 | 67
  At Month 19: Strongly agree | 17 | 30
  At Month 19: Agree | 13 | 21
  At Month 19: Neither agree or Disagree | 6 | 11
  At Month 19: Disagree | 0 | 4
  At Month 19: Strongly disagree | 0 | 1
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21: Strongly agree | 17 | 27
  At Month 21: Agree | 15 | 29
  At Month 21: Neither agree or Disagree | 6 | 6
  At Month 21: Disagree | 0 | 3
  At Month 21: Strongly disagree | 0 | 0
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24: Strongly agree | 16 | 28
  At Month 24: Agree | 19 | 25
  At Month 24: Neither agree or Disagree | 3 | 9
  At Month 24: Disagree | 1 | 2
  At Month 24: Strongly disagree | 0 | 1

17. Secondary Outcome: Subject Satisfaction: Would You Recommend the Treatment to a Friend?
Description: A subject satisfaction question with responses Yes or No.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 67
Participants
  At Month 19: number analyzed (Participants) | 36 | 67
  At Month 19: Yes | 34 | 56
  At Month 19: No | 2 | 11
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21: Yes | 35 | 58
  At Month 21: No | 3 | 7
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24: Yes | 35 | 55
  At Month 24: No | 4 | 10

18. Secondary Outcome: Subject Satisfaction: Would You do the Treatment Again?
Description: A subject satisfaction question with responses Yes or No.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 67
Participants
  At Month 19: number analyzed (Participants) | 36 | 67
  At Month 19: Yes | 31 | 55
  At Month 19: No | 5 | 12
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21: Yes | 32 | 58
  At Month 21: No | 6 | 7
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24: Yes | 34 | 55
  At Month 24: No | 5 | 10

19. Secondary Outcome: Change From Baseline in Satisfaction With Cheeks FACE-Q™ Questionnaire Rasch-transformed Total Scores
Description: The participant assessed satisfaction using the 5 questions on the FACE-Q: Satisfaction with Cheeks Appearance questionnaire measured on a 4-point scale. The responses to the items were converted to a 100-point Rasch transformed total score with 0 (worst) to 100 (best). Higher scores indicate higher satisfaction. A negative change from baseline indicates less improvement.
Time Frame: Baseline, Months 19, 21 and 24 (4 weeks is defined as one month in the study / study follow up windows for certain visits were +/- 2 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 67
score on a scale
  At Month 19: number analyzed (Participants) | 36 | 67
  At Month 19 | 42.9 (29.73) | 34.9 (37.0)
  At Month 21: number analyzed (Participants) | 38 | 65
  At Month 21 | 44 (28.41) | 38.7 (27.98)
  At Month 24: number analyzed (Participants) | 39 | 65
  At Month 24 | 45.3 (32.91) | 36.8 (30.69)

20. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs were defined as AEs with a start date on or after the first dose of investigational product or a start date before the date of the first dose of investigational product that increased in severity or after the date of the first dose. A SAE was any untoward medical occurrence (whether considered to be related to investigational product or not) that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital abnormality/birth defect, and was an important.
  medical event. TEAEs included both serious and non-serious TEAEs.
Time Frame: From start of study drug administration up to end of the study (up to Month 24) (4 weeks is defined as one month in the study / study follow up windows for certain visits were +/- 2 weeks)
Population: The extension population included all participants entering the extension study. (4 weeks is defined as one month in the study / study follow up windows for certain visits were +/- 2 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
Number analyzed (Participants) | 39 | 72
Participants
  TEAEs | 17 | 15
  Serious TEAEs | 0 | 1

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to end of the study (up to Month 24)
Description: The extension population included all participants entering the extension study.
Arm/Group | Group A: Sculptra Aesthetic | Group B: No Treatment
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/39 | 1/72
Other Adverse Events (participants affected / at risk) | 11/39 | 4/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Sculptra Aesthetic (N=39) | Group B: No Treatment (N=72)
COVID-19 pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Sculptra Aesthetic (N=39) | Group B: No Treatment (N=72)
Injection site bruising (General disorders) | 5 | 0
Injection site pain (General disorders) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
COVID-19 (Infections and infestations) | 0 | 4
Postmenopause (Social circumstances) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT04595331/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT04595331/SAP_001.pdf